CLINICAL TRIAL: NCT03832933
Title: Comparing High and Normal Protein Diets for the Dietary Remission of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, James O. Hill, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300002928
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Type 2; Obesity; Diet Modification
Keywords: weight loss; dietary protein
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Loss | interventions — Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Protein Diet (Experimental)
  Interventions: Behavioral: High Protein Diet
- Standard Protein Diet (Active Comparator)
  Interventions: Behavioral: Standard Protein Diet

INTERVENTIONS:
Behavioral: High Protein Diet — 16 week weight loss and 36 weight loss maintenance intervention. Approximate macronutrient distributions (carbohydrate:protein:fat) will be 32%:40%:28%.
  Arms: High Protein Diet
Behavioral: Standard Protein Diet — 16 week weight loss and 36 weight loss maintenance intervention. Approximate macronutrient distributions (carbohydrate:protein:fat) will be 53%:21%:25%.
  Arms: Standard Protein Diet

SUMMARY:
The purpose of this study is to examine the impact of high protein (HP) vs. normal protein (NP) diets on weight loss, loss of fat free mass (FFM), and remission of type 2 diabetes (T2D) in individuals with T2D. Both diet groups will receive dietary and physical activity guidance through a group-based weight loss program, State of Slim (SOS). The central hypothesis is that the HP diet (with ≥4 weekly servings of lean beef) will lead to greater remission of T2D vs. a NP diet by 1) producing greater weight loss and limiting weight regain and 2) preferentially reducing fat mass while preserving FFM.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥18 years
* T2D diagnosis within previous 6 years (documented physician diagnosis, use of antidiabetic medication, fasting glucose ≥126 mg/dl, and/or HbA1c ≥6.5%)
* BMI of ≥27 kg/m2
* Weight stable (±3kg in the last 3 months)
* Participants using GLP-1 agonists or SLGT-inhibitors must be on a stable (≥3 months) medication dosage and not be planning to change medication dosage
* Willing and able to participate in a weekly group class for the first 16 weeks of the study, bi-weekly classes for the remainder of the study, and willing to participate in 4 study visits over the 52 week study period.

Exclusion Criteria:

* HbA1c concentration of ≥12%.
* Pregnant or lactating within the past 6 months or trying to become pregnant.
* Individuals following a vegetarian/vegan only diet
* Food allergies (to red meats or other common protein sources)
* Using exogenous insulin for T2D management
* Taking other medications that could cause weight loss or weight gain (such as steroids, tricyclic antidepressants, chemotherapy, antipsychotics, prescribed or OTC weight loss agents). Oral contraceptives can be used as long as subject agrees to not change use of these during the study. Vitamins and minerals that do not have a weight effect are allowed as long as use is continued without change during the study.
* Current alcohol or drug abuse or dependence (Subjects who have quit smoking in the last 6 months will be excluded. Smokers whose smoking habits have been stable for the last 6 months and which remain stable during the study can be included).
* Current Eating disorder (anorexia or bulimia)
* Any medical condition for which following a high protein diet and/or 70 minutes of exercise daily would be inadvisable.
* Untreated or unstable hypothyroidism. Thyroid medications must be stable for at least 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Change in body weight by weight scale | Baseline to 16 weeks
  Participant body weights will be measured on a kg scale
Change in body weight by weight scale | Baseline to 52 weeks
  Participant body weights will be measured on a kg scale

SECONDARY OUTCOMES:
Change in T2D diagnosis criteria | Baseline to 52 weeks.
  T2D diagnosis will be determined according to American Diabetes Association criteria, which includes fasting glucose <126 mg/dL or hemoglobin A1c <6.5%.
Change in % body fat | Baseline to 16 weeks
  Participant body fat will be measured by dual x-ray absorptiometry (DXA), which is the gold standard for measuring body composition.
Change in % body fat | Baseline to 52 weeks.
  Participant body fat will be measured by dual x-ray absorptiometry (DXA), which is the gold standard for measuring body composition.
Change in % fat free mass (FFM) | Baseline to 16 weeks.
  Participant FFM will be measured by dual x-ray absorptiometry (DXA), which is the gold standard for measuring body composition.
Change in % FFM | Baseline to 52 weeks.
  Participant FFM will be measured by dual x-ray absorptiometry (DXA), which is the gold standard for measuring body composition.

CONTACTS AND LOCATIONS:
Overall Officials: James Hill, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clina JG, Sayer RD, Pan Z, Cohen CW, McDermott MT, Catenacci VA, Wyatt HR, Hill JO. High- and normal-protein diets improve body composition and glucose control in adults with type 2 diabetes: a randomized trial. Obesity (Silver Spring). 2023 Aug;31(8):2021-2030. doi: 10.1002/oby.23815. PMID 37475689